CLINICAL TRIAL: NCT02650180
Title: Usability Study for SOBERLINK System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soberlink Healthcare LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: USPROT 2015-001
Record Dates: First submitted 2015-12-29; First posted 2016-01-08 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Alcoholism; Alcohol Dependence
Keywords: Rehabilitation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Soberlink Cellular Device (Other): Soberlink Cellular Device: a Breath Alcohol Analyzer
  Interventions: Device: Soberlink Cellular Device

INTERVENTIONS:
Device: Soberlink Cellular Device — Alcohol Breath Analyzer

SUMMARY:
The Soberlink Cellular device, in its original packaging, along with the QuickStart guide will be provided to the end user in a simulated home use environment or by Rx in clinic. The patient labeling will be in the format intended for distribution.

Ten (10) Rx subjects will be provided instruction for use in clinic for the Soberlink Cellular device while an additional ten (10) Rx subjects will be provided instruction for use in clinic for the Soberlink Cellular device and Sober Sky web portal. An additional ten (10) simulated home use subjects will be provided instruction for use for the Soberlink Cellular device while an additional ten (10) simulated home use subjects will be provided instruction for use in clinic for the Soberlink Cellular device and Sober Sky web portal. All subjects will be provided with a post-test questionnaire on how to operate the device.

The post-test questionnaire will collect information regarding device use. The device's use will be compared with identified risks to determine if the percentage of failures is within the study protocol success criteria. Additionally, measurable usability criteria for specific, critical steps will be evaluated.

DETAILED DESCRIPTION:
Forty (40) subjects identified as potential end users of the device will be recruited to the study and screened according to the study inclusion and exclusion criteria. Subjects will be asked to sign informed consent. The Soberlink Cellular device, in its original packaging, along with the QuickStart guide will be provided to the patient in a simulated home-use environment and Rx clinical setting. The patient labeling will be in the format intended for distribution.

Ten (10) Rx subjects will be provided instruction for use in clinic for the Soberlink Cellular device while an additional ten (10) Rx subjects will be provided instruction for use in clinic for the Soberlink Cellular device and Sober Sky web portal. An additional ten (10) simulated home use subjects will be provided instruction for use for the Soberlink Cellular device while an additional ten (10) simulated home use subjects will be provided instruction for use in clinic for the Soberlink Cellular device and Sober Sky web portal. All subjects will be provided with a post-test questionnaire on how to operate the device.

The post-test questionnaire will collect information regarding device use. The device's use will be compared with identified risks to determine if the percentage of failures is within the study protocol success criteria. Additionally, measurable usability criteria for specific, critical steps will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18-99 years old in a clinical setting under the care of a healthcare provider.
* Male and female participants between the ages of 18-99 years old in an over-the-counter setting (home use setting).

Exclusion Criteria:

* Participants with lung disease unable to exhale for 4 seconds.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Operating the Soberlink Cellular device | 30 minutes
  Using the device with the Quick Start Guide, all 40 subjects tested are expected to be able to complete device related tasks, including starting the application, operating the Soberlink Cellular device and obtaining a breath reading and recording the results, in a timeframe of up to 30 minutes and with minimal attempts to ask for assistance; and using the device and the Quick Start Guide. Considering that the Soberlink Cellular device is a low risk device, and the probability of an occurrence and the severity of a failure are low, a success rate of 100% potential end user subjects passing may be considered acceptable for the over the counter use of the device. Any failures to complete the device related tasks and/or self-exclude from use of the device must be explained.

SECONDARY OUTCOMES:
Participants' level of success in recollecting tasks related to the use of the Soberlink Cellular device and application. | 30 minutes
  Numerical ratings describing the participants' level of success in recollecting tasks will be collected through user post-test questionnaire responses and will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Costa, BA, Study Director — Soberlink Healthcare LLC
Locations (3):
- United States (3):
  - Private Practice, Fullerton, California
  - Addiction Alternatives, Los Angeles, California
  - Hazelden Betty Ford, Center City, Minnesota

IPD SHARING:
Plan to Share IPD: No